CLINICAL TRIAL: NCT05010239
Title: The Immediate Effect of Mindfulness-Based Supportive Therapy (MBST) vs Supportive Listening on Palliating Suffering in Palliative Care Cancer Patients: A Randomised Controlled Trial
Brief Title: The Immediate Effect of Mindfulness-Based Supportive Therapy on Palliating Suffering in Palliative Care Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Malaysia Sarawak (Other)
Collaborators: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202089-8970
Record Dates: First submitted 2021-08-10; First posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Cancer; Suffering
Keywords: mindfulness; supportive; cancer; suffering; palliative
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel group, single-blinded, randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Patients in the intervention group will receive a 30-minute MBST session by a palliative care physician trained in mindfulness practice. The MBST consists of a session that involves interviewing patients with open-ended questions on suffering experiences. During the session, the practitioner will practice mindful breathing simultaneously while listening to patients. The practitioner will acknowledge the distress of patients when it is appropriate, but without losing their attention on mindful breathing. Outcomes will be measured at baseline and at minute 30.
  Interventions: Other: 30-minute Mindfulness-Based Supportive Therapy
- Control group (Placebo Comparator): Patients in the control group will receive a 30-minute supportive listening session by a palliative care physician who has no experience in mindfulness practice. The session involves interviewing patients with the same open-ended questions on suffering experiences. The practitioner will acknowledge the distress of patients when it is appropriate. Outcomes will be measured at baseline and at minute 30.
  Interventions: Other: 30-minute supportive listening

INTERVENTIONS:
Other: 30-minute Mindfulness-Based Supportive Therapy — The MBST consists of a session that involves interviewing patients with open-ended questions on suffering experiences. During the session, the practitioner will practice mindful breathing simultaneously while listening to patients. The practitioner will acknowledge the distress of patients when it is appropriate, but without losing their attention on mindful breathing.
  Arms: Intervention group
Other: 30-minute supportive listening — Patients in the control group will receive a 30-minute supportive listening session by a palliative care physician who has no experience in mindfulness practice. The session involves interviewing patients with the same open-ended questions on suffering experiences. The practitioner will acknowledge the distress of patients when it is appropriate. Outcomes will be measured at baseline and at minute 30.
  Arms: Control group

SUMMARY:
The was a parallel group, single-blinded, randomized controlled trial comparing the effectiveness of 30-minute mindfulness-based supportive therapy versus supportive listening in reducing suffering among patients with cancer. This study was conducted in the University Malaya Medical Centre, from 1st august 2020 to 31 December 2020.

DETAILED DESCRIPTION:
This study was conducted in the University Malaya Medical Centre. The study design was a parallel-group, single-blinded, randomized controlled trial. The trial will be registered at the Clinical Trials registry and was conducted in accordance to the Declaration of Helsinki. The investigators recruited patients by screening patients under the care of the palliative care team at University Malaya Medical Centre. Patients fulfilling the inclusion and exclusion criteria will be approached and included in the study if give informed consent to participate.

Inclusion criteria:

* Stage III and IV cancer patients aged 18 years and above
* The overall suffering score of 4/10 and above based on The Suffering Pictogram

Exclusion criteria:

* Patients who are confused based on The Confusion Assessment scoring
* Patients who are non-communicative verbally
* Patients with psychiatric illness

Patients who were eligible were informed about the nature of the study. The study was voluntary and patients could withdraw from the study at any time. Patients who were interested to participate was randomly allocated to either the intervention group (MBST) or the control group (supportive listening) based on computer generated random numbers. Allocation concealment will be performed using sealed envelopes.

Patients in the intervention group received a 30-minute MBST session by a palliative care physician trained in mindfulness practice. The MBST consisted of a session that involvesd interviewing patients with open-ended questions on suffering experiences. During the session, the practitioner practiced mindful breathing simultaneously while listening to patients. The practitioner acknowledged the distress of patients when it was appropriate, but without losing their attention on mindful breathing.

Patients in the control group received a 30-minute supportive listening session by a palliative care physician who has no experience in mindfulness practice. The session involves interviewing patients with the same open-ended questions on suffering experiences. The practitioner acknowledged the distress of patients when it was appropriate. Outcomes will be measured at baseline and at minute 30.

Primary outcomes (patients): Suffering was measured using the Suffering Pictogram. It is a brief and validated instrument used to measure the experience of suffering in palliative care. Patients were required to rate overall suffering at the centre of the pictogram with a numerical scale of 0 to 10 (0 = no suffering, 10 = worst possible suffering). The pictogram contains eight items rated on a Likert scale - discomfort, worry, fear, anger, sadness, hopelessness, difficulty in acceptance and emptiness. The total suffering score of the eight items ranged from 0 to 32, with higher score reflecting more suffering.

Psychological distress was examined using the Hospital Anxiety and Depression Scale (HADS). The HADS consisted of 14 items rated on a Likert scale yielding a score of total score (0-42), an anxiety score (0-21) and a depression score (0-21), with higher score reflecting higher distress.

Quality of life (QOL) was assessed by the Functional Assessment of Chronic Illness Therapy (FACIT-Sp). It contained 39 items (range from 0 to 4, with higher scores reflecting higher QOL) forming an overall total score and five subscales scores: physical, social, emotional, functional and spiritual.

Patient's perception of practitioner empathic engagement was measured with the Jefferson Scale of Patient's Perceptions of Physician Empathy. It was a 5-item instrument (range from 1 to 5, with higher scores reflecting a greater degree of physician's empathy).

Secondary outcomes (practitioners): Secondary outcomes were measured by the Perceived Stress Scale (PSS) and the Frieburg Mindfulness Inventory (FMI).

ELIGIBILITY:
Inclusion Criteria:

* Stage III and IV cancer patients aged 18 years and above
* The overall suffering score of 4/10 and above based on The Suffering Pictogram

Exclusion Criteria:

* Patients who are confused based on The Confusion Assessment scoring (CAM)
* Patients who are non-communicative verbally
* Patients with psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Suffering measured using the Suffering Pictogram. | 30-minute
  Suffering pictogram is in numerical scale of 0 to 10 (0 = no suffering, 10 = worst possible suffering). The pictogram contains eight items rated on a Likert scale - discomfort, worry, fear, anger, sadness, hopelessness, difficulty in acceptance and emptiness. The total suffering score of the eight items ranges from 0 to 32, with higher score reflecting more suffering.
Psychological distress examined using the Hospital Anxiety and Depression Scale. | 30-minute
  Hospital Anxiety and Depression Scale consists of 14 items rated on a Likert scale yielding a score of total score (0-42), an anxiety score (0-21) and a depression score (0-21), with higher score reflecting higher distress.
Quality of life assessed by the Functional Assessment of Chronic Illness Therapy. | 30-minute
  Functional Assessment of Chronic Illness Therapy, contains 39 items (range from 0 to 4, with higher scores reflecting higher quality of life) forming an overall total score and five subscales scores: physical, social, emotional, functional and spiritual.
Patient's perception of practitioner empathic engagement measured with the Jefferson Scale of Patient's Perceptions of Physician Empathy | 30-minute
  Jefferson Scale of Patient's Perceptions of Physician Empathy is a 5-item instrument (range from 1 to 5, with higher scores reflecting a greater degree of physician's empathy).

SECONDARY OUTCOMES:
Perception of stress measured by Perceived Stress Scale | 30-minute
  Perceived Stress Scale has 10 items, each range 0 - never to 4 - very often. The total score is 40, with higher score indicates more perceive stress.
Mindfulness measured by Frieburg Mindfulness Inventory | 30-minute
  Frieburg Mindfulness Inventory has 14 items, from 1 (rarely) to 4 (always). The higher the total score, the higher the mindfulness.

CONTACTS AND LOCATIONS:
Overall Officials: Chee-Shee Chai, MD, Study Director — Faculty of Medicine and Health Science, University Malaysia Sarawak
Locations (1):
- University Malaya Medical Center, Kuala Lumpur, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No
The data can be requested from the primary investigators. The data cannot upload to the public repository due to restrictions from the ethics committee.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/39/NCT05010239/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/39/NCT05010239/ICF_001.pdf